CLINICAL TRIAL: NCT01962285
Title: Neuronal Inertia´s Effect on Pharmacological Behavior Representation of Propofol
Brief Title: Neuronal Inertia in Propofol Anesthesia
Acronym: INERTIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad del Desarrollo (Other)
Responsible Party: Principal Investigator, Pablo Sepulveda, Médico Cirujano, Universidad del Desarrollo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: INERTIA
Record Dates: First submitted 2013-10-09; First posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: General Anesthesia; Propofol Pharmacodynamics; Propofol Target Controlled Infusion; Loss of Consciousness and Recovery of Consciousness; Propofol Plasma Concentration
Keywords: neuronal inertia; loss of consciousness; propofol pharmacodynamics; Bispectral index; anesthesia, general/pharmacology
MeSH Terms: conditions — Unconsciousness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- propofol slow infusion (Experimental): (healthy volunteers, non invasive monitoring and O2 supply via nasal cannula) Target controlled infusion of propofol using Schnider´s pharmacokinetic parameters in a slow, stepped fashion. beginning at Cp 0.5 mcg/ml and increasing in 0.5 mcg/ml every 7 minutes until LOC occurred, then a prolonged step of 14 minutes (2 samples), increase 2 steps further and then decrease in 0.5 mcg/ml steps until ROC and a 7 minute registry after ROC.
  Blood sampling for propofol plasma level every 7 minutes (at the end of each step, allowing for pseudo-equilibrium condition.
  32 channel-EEg and BIS continuous monitoring
  Interventions: Drug: propofol targel controlled infusion

INTERVENTIONS:
Drug: propofol targel controlled infusion — slow stepped propofol target controlled infusion using Schinider´s pharmacokinetic parameters seriated venous blood sampling
  Other Names: propofol TCI

SUMMARY:
Loss and recovery of consciousness during propofol anesthesia seem to be mediated by different mechanisms beyond the actual effect-site concentration of anesthetic drug. This eventual difference between dose response curves for loss of consciousness (LOC) and for recovery of consciousness (ROC) beyond hysteresis has received the name of neuronal inertia. We performed a volunteer-study comparing LOC and ROC curves during a slow, steady-sate, stepped target controlled infusion of Propofol. Our hypothesis is that, at steady-state conditions between plasma an effect-site concentration, there is still going to exist a difference between LOC and ROC, demonstrating the existence of neuronal inertia.

DETAILED DESCRIPTION:
Loss and recovery of consciousness during propofol anesthesia seem to be mediated by different mechanisms beyond the actual effect-site concentration of anesthetic drug. This eventual difference between dose response curves for loss of consciousness (LOC) and for recovery of consciousness (ROC) beyond hysteresis has received the name of neuronal inertia. We performed a volunteer-study comparing LOC and ROC curves, during a slow, steady-sate, stepped target controlled infusion of Propofol using Schnider's pharmacologic model. Our hypothesis is that, at steady-state conditions between plasma an effect-site concentration, there is still going to exist a difference between LOC and ROC, demonstrating the existence of neuronal inertia.

ELIGIBILITY:
Inclusion Criteria:

* american society of anesthesiologists status I or II age >18 years fasted at least 8 hours BMI<30

Exclusion Criteria:

* any known adverse reaction to propofol administration soy or egg-protein allergy psychotropic use (illegal of medically indicated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-08; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
plasma-equilibrated effect site concentration of propofol at LOC and ROC (mcg/ml) | 2 hours (during slow steady-state concentration propofol infusion)
  determination of plasma concentration of PROPOFOL at the time of Loss of Consciousness and the time of recovery of consciousness during the 7-minute step infusion.
  Provided it is a slow increasing infusion we assume a pseudo-equilibrium state between plasma and effect site.
  the existence of a difference between these two values will support the hypothesis of neuronal inertia

SECONDARY OUTCOMES:
Bispectral Index (BIS) al LOC and ROC | 2 hours (during slow increasing TCI (Target controlled Infusion) of PROPOFOL
  we measured the BISPECTRAL INDEX all through the protocol: from previous to start the infusion until 7 minutes after recovery of consciousness. values of BIS at LOC and ROC will be compared.
  a potential difference found between those two values supports the theory thas LOC and ROC reflects different neuronal processes Other clinically relevant endpoints (loss of palpebral reflex, onset of amnesia) will be registered in order to build the pharmacodynamic loop.
Pharmacodynamic curve for propofol. | 2 hours
  plasma concentration of PROPOFOL (mcg/ml) at other clinically relevant endpoints (amnesia onset, loss of palpebral reflex, etc...) will be determined in order to build a pharmacodynamic curve,
PROPOFOL effect site concentration during infusion | 2 hours
  plasma concentration of PROPOFOL (mcg/ml) from venous blood samples will be determinated every 7 minutes, that means at the end of each TCI step. assuming the 7-minute step gave enough time to reach a pseudo-equilibrium state, we consider the results comparable to effect site concentration.

OTHER OUTCOMES:
performance of Schnider´s pharmacokinetic parameters in a slow infusion | 2 hours
  to compare plasma (and effect site) Propofol concentration predicted by the model with measured values thus evaluating model´s performance. Median performance error (MDPE) and median absolute performance error (MDAPE), divergence and other often reported parameters will be determinated.
Electroencephalographic behavior at LOC and ROC during Propofol infusion | 2 hours (during propofol infusion)
  spectral analisis of 32-channel EEG during infusion. a specified time-frame around those two events (i.e.: 14 minutes) will be reconstructed in images and analyzed. cortical areas with enhanced activity and how do this activity changes during loss of consciousness and the recovery of it will be evaluated with a mathematical model in order two determine wether those events correspond with two different processes instead of a bidirectional single one.

CONTACTS AND LOCATIONS:
Overall Officials: pablo sepulveda, anesthesiologist, Principal Investigator — Universidad del Desarrollo
Locations (1):
- Clinica Alemana de Santiago, Santiago, Santiago Metropolitan, Chile